CLINICAL TRIAL: NCT00839020
Title: Comparison of a Minimally Invasive and a Conventional Approach in Computer Assisted Total Knee Arthroplasty.
Brief Title: Minimally Invasive Versus Conventional Approaches in Navigated Total Knee Arthroplasty (TKA)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Number of patients willing to participate in the study too low
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIOS-TKR
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis
Keywords: Surgical Procedures, Minimally Invasive; Range of Motion; Articular Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Navigated total knee arthroplasty with a minimally invasive approach
  Interventions: Procedure: Navigated TKA with a minimally invasive approach
- 2 (Active Comparator): Navigated total knee arthroplasty with a conventional approach
  Interventions: Procedure: Navigated TKA with a conventional approach

INTERVENTIONS:
Procedure: Navigated TKA with a minimally invasive approach — Navigated total knee arthroplasty with a minimally invasive approach
  Other Names: Navigated MIS TKA
  Arms: 1
Procedure: Navigated TKA with a conventional approach — A navigated total knee arthroplasty is performed using the Orthopilot navigation system. A conventional approach is performed
  Other Names: Navigated TKA with conventional approach
  Arms: 2

SUMMARY:
50 patients are randomized to two groups who receive a navigated knee prosthesis. Aim of the study is a comparison between a minimally invasive and a conventional approach. In both groups OrthoPilot computer assisted-navigation will be used. Pain intensity as well as concomitant pain medication are monitored during the first 20 postoperative days and will be compared for the two groups. Various scores are surveyed.

DETAILED DESCRIPTION:
Accuracy of implant positioning and reconstruction of the mechanical leg axis are major requirements for achieving good long-term results in total knee arthroplasty (TKA). A minimally invasive approach might compromise the accuracy due to lacking intraoperative oversight. The purpose of this study is to compare a minimally invasive TKA approach that was performed under control of a navigation system with a standard navigated approach, with respect to patient pain and range of motion.

All patients receive a Columbus knee prosthesis and in both groups an OrthoPilot navigation system is used to control the alignment. Pain intensity using the Visual Analogue Scale (VAS) and concomitant pain medication intake are documented daily during the first 20 days after operation. As long as the patient is hospitalized the Range of Motion will also be documented daily. Knee society score, oxford score, as well as the WOMAC score are monitored pre- and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective TKA
* agreement to participate in this study

Exclusion Criteria:

* Body Mass Index (BMI)>40kg/m²
* varus or valgus deformity >20°
* Range of Motion (ROM) <75° flexion/extension
* concomitant diseases like: rheumatoid arthritis osteoporosis intake of cortisone diabetes former operations on the concerned knee
* infections in the operated joint during the follow-up period
* Thromboses during the follow-up period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity using the Visual Analogue Scale (VAS) regarding concomitant pain medication intake. | daily measurements for 20 postoperative days

SECONDARY OUTCOMES:
Range of Motion (ROM) | daily measurements during hospital stay
Knee Society Score (KSS) | preop, postop
Oxford Knee Score (OKS) | preop, postop
WOMAC-Score | preop, postop

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lampe, MD, Principal Investigator — Schön Kliniken Klinikum Eilbek
Locations (1):
- Frank Lampe, MD, Hamburg, Germany